CLINICAL TRIAL: NCT00292409
Title: A Prospective Open-Label Study of Aripiprazole in the Management of Patients With Schizophrenia in General Psychiatric Practices
Brief Title: A Study of Aripiprazole in Patients With Schizophrenia in General Psychiatric Practices
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CN138-125
Record Dates: First submitted 2005-09-12; First posted 2006-02-16 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia and Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this clinical research study is to evaluate the overall effectiveness of 8 week of aripiprazole treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder being treated as outpatients,no response to past antipsychotic treatment and patients who symptoms are notoptimally controlled defined as CGI- S<7

Exclusion Criteria:

* pregnant or breastfeeding,patients at risk for committing suicide,diagnosis of mood disorders, delirium, dementia and other cognitive disorders,patients treatment resistant to otherantipyschotic medications and treatment with a long acting psychotic in which the last dose was within 3 months of treatment phase

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement at endpoint

SECONDARY OUTCOMES:
Clinical Global Impression scale
Investigator's Assessment Questionnaire
Patient preference of medication at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb